CLINICAL TRIAL: NCT01628991
Title: Comparison of the Effect of Vaginal Cones and Behavioral Intervention Program on Urinary Stress Incontinence in Women
Brief Title: Behavioral Intervention Program and Vaginal Cones on SUI
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Mashhad University of Medical Sciences (Other)
Responsible Party: Principal Investigator, nahid golmakani, Faculty member,MSc of Midwifery, Mashhad University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: clinical trial
Record Dates: First submitted 2012-06-17; First posted 2012-06-27 (Estimated); Last update posted 2012-06-27 (Estimated); Status verified 2012-06

CONDITIONS: Stress Urinary Incontinence
Keywords: Behavioral Intervention Program; Vaginal Cones; Stress Urinary Incontinence; treatment; Women
MeSH Terms: conditions — Urinary Incontinence, Stress | interventions — Exercise Therapy; Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- behavioural intervention (Experimental): Recieving interventional behavioural program
  Interventions: Behavioral: behavioural program
- vaginal cone (Experimental): intravaginal device insertion(vaginal cone)
  Interventions: Device: Iranian version of vaginal cones

INTERVENTIONS:
Behavioral: behavioural program — interventional behavioural program
  Other Names: bladder training program, exercise therapy
  Arms: behavioural intervention
Device: Iranian version of vaginal cones — intravaginal device(vaginal cone) for promote the pelvic floor exercises
  Other Names: intravaginal cones with different weights,Physical Therapy
  Arms: vaginal cone

SUMMARY:
This study is a single blind randomized clinical trial to compare the efficacy of a behavioral intervention program versus vaginal cones on Stress Urinary Incontinence (SUI).

DETAILED DESCRIPTION:
Detailed Description: In this single-blind randomized clinical trial, 60 women aged 25-65 yrs with stress urinary incontinence were randomly divided in two groups by blocked randomization method; behavioral intervention program (n=30) and insertion vaginal device,vaginal cones (n=30). Women in behavioral intervention group were instructed for pelvic floor exercise and bladder control strategies. Other group was allocated to use vaginal cones. They were treated for 12 weeks and followed up every 2 weeks. The subjective changes in severity of SUI were measured using a Detection SUI Severity Questionnaire and leakage index and 3-day urinary dairy. The objective changes were measured by pad test. These two groups were then compared according to the scores of special questionnaires for quality of life, strength of pelvic floor muscles, capability to participate in social activities, severity of urinary incontinence, and the number of involuntary urine passage, taken before, and after 1 and 3 months after finishing interventions. Data analysis will be done through descriptive and perceptive statistical methods by using SPSS.

ELIGIBILITY:
Inclusion Criteria:

* symptoms of SUI , at least three episodes of stress incontinence per week
* Age 25-65
* body mass index (BMI) ≤ 30 kg/m2
* physical health

Exclusion Criteria:

* chronic degenerative diseases affected on muscular and nerve tissues
* vulvovaginitis, atrophic vaginitis,
* pregnancy
* active or recurrent urinary tract infections
* advanced genital prolepses
* patients with cardiac pacemakers

Ages: 25 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2008-04; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
severity of Stress Urinary Incontinence | three months

SECONDARY OUTCOMES:
Quality of life | three months

CONTACTS AND LOCATIONS:
Overall Officials: Nahid golmakani, M.Sc., Study Director — Mashhad university of medical science, faculty of nursing and midwifery, Mashhad, Iran; Nayereh khadem, M.D., Study Chair — Mashhad university of medical science, Mashhad, Iran; Arezoo Arabipoor, M.Sc., Principal Investigator — Mashhad university of science, faculty of nursing and midwifery, Mashhad, Iran
Locations (1):
- Mashhad university of medical science, Mashhad, Iran